CLINICAL TRIAL: NCT01700452
Title: Clinical Study of BioView Target -FISH Lung Cancer Detection Test
Brief Title: Diagnostic Study for Lung Cancer Detection Test
Status: Completed | Type: Observational
Sponsor: Bioview, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LCD Test 17Jul2012; Revision 3 (Other: BioView, Inc.)
Record Dates: First submitted 2012-09-10; First posted 2012-10-04 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Pulmonary nodules; FISH Test
MeSH Terms: conditions — Lung Neoplasms; Multiple Pulmonary Nodules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sputum specimens, fixed and stained for diagnostic testing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients suspected of having lung cancer: Subjects presenting with 0.8 - 3 cm solitary pulmonary nodules with high probability for malignance. The subject must be scheduled for a lung biopsy procedure to determine clinical diagnosis.

SUMMARY:
Early detection of lung cancer and early removal of the cancer nodules facilitates the diagnosis and treatment. However, not all nodules are malignant. Currently the standard method to diagnose lung cancer is to remove any suspicious nodules from the lung in a surgical procedure.

This study is being conducted to evaluate the performance of a laboratory test to detect changes in lung cells that might be an early indicator of lung cancer. The test uses mucus (sputum) which is collected in a non-invasive method. This study will compare the results of the lung biopsy with the laboratory test to determine if the test can detect cancer or the lack of cancer.

The laboratory test will not be shared with the treating physician or the patient as the current standard for lung cancer diagnosis is a biopsy. Approximately 330 patients will be enrolled in the study. There is one visit involved and includes the collection of a sputum specimen by coughing into a cup. The medical records of patients who are negative for cancer by biopsy will be reviewed for 2 years to detect any changes in diagnosis.

DETAILED DESCRIPTION:
This study is being conducted to evaluate the performance of a laboratory test to detect changes in lung cells that might be an early indicator of lung cancer. The test uses mucus (sputum) which is collected in a non-invasive method. This study will compare the results of the lung biopsy with the laboratory test to determine if the test can detect cancer or the lack of cancer.

The laboratory test will not be shared with the treating physician or the patient as the current standard for lung cancer diagnosis is a biopsy. Approximately 330 patients will be enrolled in the study. There is one visit involved and includes the collection of a sputum specimen by coughing into a cup. The medical records of patients who are negative for cancer by biopsy will be reviewed for 2 years to detect any changes in diagnosis.

The results of the test will not be provided to the subject, the investigator and will not be used to diagnose or treat the subject.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with 0.8-3 cm solitary pulmonary nodules with high probability for malignancy
* Candidate is scheduled to undergo lung biopsy procedure to determine clinical diagnosis, such as Bronchoscope biopsy, Electromagnetic Navigation Bronchoscopy, fiber optic Bronchoscopy, Needle biopsy, CT guided, Percutaneous Transthoracic Needle biopsy, Transthoracic Needle Biopsy, Open biopsy for Diagnostic Resection or Video-Assisted Thorascopic Surgery.
* Candidate who is capable of undergoing sputum induction.
* Ability to understand the investigational nature of the study and sign the informed consent.

Exclusion Criteria:

* Subjects who pose a high clinical risk for diagnostic bronchoscopy or transthoracic biopsy for definitive diagnosis.
* Subjects already diagnosed with lung cancer, or previously treated for lung cancer.
* Subjects who experienced pneumonia within last 12 weeks.
* Subjects who experienced an acute respiratory infection within the last 2 weeks
* Cases without sufficient documentation of diagnosis or follow-up will not be included.
* Treatment for, or evidence of any cancer other than nonmelanoma skin cancer or carcinoma in situ within the last 3 years.
* Subject who lack the capacity to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects will be selected from pulmonary clinics and physician's practice in community hospital settings.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2012-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Determination of concordance of the Target-Fish LCD Test and diagnosis by biopsy | 2 weeks following sputum collection
  Subjects suspected of having of having lung cancer and who are to undergo biopsy will undergo sputum sampling. The sputum will be assayed using the BioView test kit. Biopsy results will be compared with the assay results, each being a dichotomous response (positive or negative for cancer by biopsy, positive or negative assay result using client-supplied cut-off). Since the assay may detect cancer before a biopsy is positive or because the sputum sampling may be more representative of the condition of the lung than just the biopsied nodule, it will be necessary to follow thte negative biopsy subjects for up to two years to either rule in or rule out lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Schwebel, PhD, Study Director — Bioview, Inc.
Locations (6):
- United States (3):
  - VA Greater Los Angeles Health System, Los Angeles, California
  - Frederick Memorial Hospital, Regional Cancer Center, Frederick, Maryland
  - St. Luke's Hospital, Bethlehem, Pennsylvania
- Israel (3):
  - Kaplan Medical Center, Rehovot
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center Thoracic Cancer Research and Detection Center, Tel Litwinsky

IPD SHARING:
Plan to Share IPD: No